CLINICAL TRIAL: NCT01821768
Title: A Prospective Randomized Trial of Sentinel Lymph Node Biopsy Versus no Additional Staging in Patients With Clinical T1-T2 N0 M0 Invasive Breast Cancer and Negative Axillary Ultrasound
Brief Title: Axillary Ultrasound With or Without Sentinel Lymph Node Biopsy in Detecting the Spread of Breast Cancer in Patients Receiving Breast Conservation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201209143
Record Dates: First submitted 2013-03-20; First posted 2013-04-01 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: No sentinal lymph node biopsy (No Intervention): Patients will receive no additional axillary surgery which is experimental.
- Arm 2: Sentinel lymph node biopsy (Active Comparator): Patients will receive standard of care sentinel lymph node biopsy
  Interventions: Procedure: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy
  Arms: Arm 2: Sentinel lymph node biopsy

SUMMARY:
This randomized clinical trial studies two different tests that are currently being used to detect the spread of breast cancer to the lymph nodes under the arm in candidates for breast conservation therapy. The two tests are sentinel lymph node biopsy (SLNB) and axillary ultrasound. The current standard of care is sentinel lymph node biopsy, which is a surgical procedure. Axillary ultrasound (AUS) may be just as good as SLNB for detecting the spread of cancer but without the surgical risks.

DETAILED DESCRIPTION:
In this prospective randomized non-inferiority study we aim to determine the utility of axillary ultrasound (AUS) as a pre-operative staging modality for patients with clinically node-negative invasive breast cancer with the hope that it will be a minimally invasive replacement for SLNB.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be female.
* Patient must be at least 18 years of age.
* Patient's clinical stage must be documented as tumor size less than 5 cm, with no palpable nodes and no evidence of metastatic disease (T1 or T2 N0 M0). For patients who will receive neoadjuvant systemic therapy, pre-treatment clinical stage should be used.
* Patient must have a negative (normal) axillary ultrasound performed at Siteman Cancer Center. Lymph nodes will be evaluated based on morphologic features. AUS wil be considered positive (abnormal)if lymph nodes are noted to be completely hypoechoic (absent hilum) or have focal hypoechoic cortical thickening/lobulation greater than 4 mm.
* Patient must have a tissue diagnosis of invasive breast carcinoma
* Patient must have Eastern Cooperative Oncology Group (ECOG) status </= 2, as documented in patient's medical record.
* Patient must be available for follow-up.
* A patient with a history of previous malignancy is eligible for this study as long as the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided that the following criteria are met (1) The patient has undergone potentially curative therapy for all prior malignancies; (2) There has been no evidence of any prior malignancies for at least five years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone); and (3) The patient is deemed by their treating physician to be at low risks for recurrence from prior malignancies.
* Patient, or the patient's legally acceptable representative, must provide a signed and dated written informed consent prior to registration and any study-related procedures.
* Patient must provide written authorization to allow the use and disclosure of their protected health information. NOTE: This may be obtained in either the study-specific informed consent or in a separate authorization form and must be obtained from the patient prior to study registration.
* Patient must be a candidate for sentinel lymph node biopsy (SLNB).

Exclusion Criteria:

* Patient in lactating (breast-feeding) or pregnant.
* Patient has concurrent invasive bilateral breast malignancies or multicentric disease.
* Patient has had previous ipsilateral axillary surgery such as excisional biopsy of lymph nodes(s), treatment of hidradenitis.
* Patient is considered poor candidate surgical candidate due to non-malignant systemic disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Regional (axillary) recurrence | 5 years from date of surgery
  The distributions of the primary endpoints and complications across two arms will be summarized using contingency tables and compared by 2-sample Chi-square test or Fisher's exact test.

SECONDARY OUTCOMES:
Disease free survival Arm 1 versus Arm 2. | At least 5 years form date of surgery to date of any disease recurrence.
  Defined as the interval between the date of registration to the date of first disease event. Kaplan-Meier product limit estimator will be used. The differences in OS and DFS between treatment arms will be compared using log-rank test.
Overall survival Arm 1 versus Arm 2 | 5 years from date of surgery
  Defined as the interval between the date of initial diagnosis until the date of death. Kaplan-Meier product limit estimator will be used. The differences in OS and DFS between treatment arms will be compared using log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Cyr, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu